CLINICAL TRIAL: NCT07406009
Title: The Psychosocial Functioning of Adults With Phenylketonuria.
Acronym: CoMet-PCU
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2025PI020
Record Dates: First submitted 2026-01-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-11

CONDITIONS: Phenylketonuria (PKU)
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient
- Relative

SUMMARY:
Current recommendations are to maintain Phe levels < 360 µmol/L throughout life (US consensus) or < 600 µmol/L from the age of 12 (European consensus). Nevertheless, these recommendations do not take into account the individuality of each PKU patient who, in reality, reacts differently to Phe levels, with some patients with high levels (> 1200 µmol/L) escaping the neurological consequences of high Phe levels without this being well understood (OJRD 2018; 13: 149. Can untreated PKU patients escape from intellectual disability? A systematic review). It is therefore unclear what blood levels of phenylalanine are required during adolescence and adulthood to maintain an optimal cognitive, emotional and neurophysiological state in individual PKU patients, depending on their personal responsiveness to Phe.

ELIGIBILITY:
Inclusion Criteria:

Patients :

* Age ≥ 18 years and < 59 years (age limit for ASEBA questionnaire)
* Person being monitored for PKU / HMP
* Relative living with the person
* Person who has received full information on the organization of the research and has not objected to the use of this data
* Compulsory membership of a social security scheme

Relatives:

* Age ≥ 18 years
* Person who has received full information on the organization of the research and has not objected to the use of this data
* Compulsory membership of a social security scheme

Exclusion Criteria:

* Refusal or linguistic, physical or psychological incapacity to to participate in the study
* Subjects under court protection
* Subjects under guardianship or curatorship

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will be offered to all adult subjects and their close relatives who know the person well as part of the follow-up for PKU at the Centre de Référence des maladies héréditaires du métabolisme at the Nancy CHRU.
  This study will be offered to a second metabolic reference center.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Total score ASEBA | single time point upon the study enrollment
  Total score ASEBA

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://depistage-neonatal.fr/wp-content/uploads/2023/01/Rapport-Activite-2021.pdf